CLINICAL TRIAL: NCT00799149
Title: Phase 4 Study Comparing the Efficacy of Etoricoxib Versus Gabapentin as Part of a Multimodal Analgesic Regimen for Ambulatory Knee Arthroscopy
Brief Title: Etoricoxib Versus Gabapentin for Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Masha Zakotski MD, Department of Anesthesiology, Meir Medical Center, Kfar Sava
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMC-045-06
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Knee Arthroscopy
Keywords: Post-operative pain; Knee arthroscopy; Gabapentin; Etoricoxib; Elective ambulatory knee arthroscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Etoricoxib; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gabapentin (Active Comparator): Gabapentin (1200 mg) administered 30-90 min before the patient entered the operating room; Subsequent doses of Gabapentin (1200 mg)were administered on the mornings (08H00) of the first, second, and third postoperative days.
  Interventions: Drug: Gabapentin, Etoricoxib, Sugar pill
- Etoricoxib (Active Comparator): Etoricoxib (120 mg)administered 30-90 min before the patient entered the operating room; Subsequent doses of etoricoxib (120 mg)were administered on the mornings (08H00) of the first, second, and third postoperative days.
  Interventions: Drug: Gabapentin, Etoricoxib, Sugar pill
- Sugar pill (Placebo Comparator): Sugar pill administered 30-90 min before the patient entered the operating room. Subsequent doses of Sugar pill were administered on the mornings (08H00) of the first, second, and third postoperative days.
  Interventions: Drug: Gabapentin, Etoricoxib, Sugar pill

INTERVENTIONS:
Drug: Gabapentin, Etoricoxib, Sugar pill — Control (Sugar pill) or gabapentin (1200 mg) or etoricoxib (120 mg) administered 30-90 min before the patient entered the operating room with a sip of water. Subsequent doses of the oral study drugs were administered on the mornings (08H00) of the first, second, and third postoperative days. .

SUMMARY:
To determine that when administered as part of a multimodal analgesic regimen, use of the new COX-2 antagonist etoricoxib (120 mg/day, per os) is more effective in improving postoperative pain management after knee arthroscopy than gabapentin (1.2 g/day, per os).

DETAILED DESCRIPTION:
Background: Post-discharge pain remains a significant problem after many ambulatory surgery procedures. Both etoricoxib and gabapentin have been used to prevent postoperative pain; however their relative efficacy in the post-discharge period is not known. We hypothesized that daily use of etoricoxib would offer advantages over gabapentin as part of a multimodal analgesic regimen in the perioperative period due to its pharmacokinetic profile.

Methods: Seventy-five healthy outpatients undergoing elective ambulatory knee arthroscopy were randomly assigned to receive identical-appearing capsules containing either a placebo, gabapentin (1.2g, or etoricoxib 120 mg, 30-90 min before skin incision and at 08H00 on the first, second, and third postoperative days. Post-discharge pain was treated with "rescue" dipyrone syrup (500 mg). Pain intensity (as assessed using a 100 visual analog scale), dipyrone usage, and the incidence of nausea and vomiting, sedation and anxiety were recorded at specific time intervals in the postoperative period. The recovery of functional activity was assessed at 96 h after surgery using a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Elective ambulatory knee arthroscopy

Exclusion Criteria:

* History of clinically-significant cardiovascular,pulmonary,hepatic,renal, neurologic, psychiatric or metabolic disease
* Patients chronically receiving pain killers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
1)Pain intensity (as assessed using a 100 visual analog scale) 2)Incidence of dipyrone usage | 96 hours post-operation

SECONDARY OUTCOMES:
The recovery of functional activity | 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel